CLINICAL TRIAL: NCT03516032
Title: Effect of Physiotherapy and Rehabilitation Program on Physical Activity Level in the Elderly Inpatient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Karapınar, PT, MSc, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15/750
Record Dates: First submitted 2018-04-04; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Hospitalism
Keywords: exercises therapy; rehabilitation; aged; inpatients
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The specific purpose of the clinical staff study not directly involved in the study is not specified in terms of not affecting the participants.
Oversight: Data Monitoring Committee: No

ARMS (2):
- walking exercises (Experimental): walking in the hospital corridor
  Interventions: Behavioral: exercises
- balance exercises (Experimental): heel rise exercises
  Interventions: Behavioral: exercises

INTERVENTIONS:
Behavioral: exercises

SUMMARY:
In inpatient older adults, decrement in their mobility and loss in their physical activity are seen in time line between their hospitalization and discharge. The aim of our study was to investigate the effect of physiotherapy and rehabilitation program on physical activity, functional skills and quality of life in elderly inpatient. A total of 124 patients who were randomized as study and control group followed by Hacettepe University Faculty of Medicine Department of Internal Medicine, Division of Geriatric Medicine were included to the study. Thirty minutes physiotherapy and rehabilitation program was applied to the patients in the study group according to their functional levels. Geriatric patients in the control group did exercises by themselves. Demographic data, cognitive functions, muscle strength, presence of comorbidity, functional mobility, physical activity, daily living activities, fear of fall, quality of life and depression status were assessed of all cases. Activities of daily living and depression status was questioned again three months later. This study evaluated the efficacy and cost effectiveness of increasing physical activity in older people during inpatient rehabilitation. These results could assist in the development of evidenced-based rehabilitation programs for this population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Mini Mental State Examination score greater than 24;
* Stayed in the hospital at least 48 hours.

Exclusion Criteria :

* Angiina pectoris, acute myocarditis, myocardial infarction story in the last 3 months,
* Pulmonary embolism and deep vein thrombosis within the last 3 months,
* Active infection,
* Malignancy and terminal disease status,
* Fracture story in the lower and upper extremities in the last three months
* Severe hearing and visual loss.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 323 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
DEMMI-De Morton Mobility Scale | 5 DAYS
  The De Morton Mobility Scale (DEMMI) was used to record the changes in mobility of the patients from admission to discharge. The score is between 0-100, and high scores indicate that mobility is better. Performance of a wide range of mobility tasks such as getting in and out of bed, standing from a chair and walking is observed and scored. The DEMMI has demonstrated reliability and validity in older adults
EQ5D-EQ-5D EuroQool Health Quality Assesment | 5 DAYS
  For quality of life assessment, we used the EuroQol- 5 Dimension (EQ-5D). The EQ-5D describes health status according to five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three levels, namely, "no problems", "some problems" and "severe problems". Besides the five dimensions, the EQ-5D consists of a visual analogue scale (VAS-5D) ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
PAIR-Physical Activity in Inpatient Rehabilitation Assessment | 5 DAYS
  Patient mobility was assessed by Physical Activity in Inpatient Rehabilitation Assessment (PAIR). PAIR was developed to allow an estimation of physical activity levels in inpatients. PAIR was to provide a cost-saving and widely available tool which is easy to implement within the rehabilitation process. This scale is scored between 0 and 7; "0" indicates that the patient is only in bed to recover, and "7" indicates that the patient can walk to the outside of the hospital to recover

SECONDARY OUTCOMES:
Katz Activities of Daily Living Scale | 5 DAYS
  The basic activities of daily living were evaluated using Katz Activities of Daily Living (ADL) Scale. It includes six categories of activities: bathing, dressing, toilet needs, transfer, continence and feeding. Each item has three response options: dependent, partially dependent or independent. A score of 6 points on the scale shows dependence, a score between 7 and 12 shows partial dependence, and a score between 13 and 18 shows independence
GDS-Geriatric Depression Scale | 10 AND 90 DAYS
  Depression statues was measured using the Geriatric Depression Scale - Short Form (GDS-15) which was developed and validated for measurement of depressive symptoms among elderly people. This scale has been widely used as a screening tool for depressive disorders in older people, with valid and reliable psychometric measures.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karapinar M, Kirdi N, Firat T. Effectiveness of supervised and functional level-based exercise program in elderly inpatients: Randomised controlled trial. Clin Rehabil. 2022 Dec;36(12):1623-1634. doi: 10.1177/02692155221116818. Epub 2022 Jul 25. PMID 35880264